CLINICAL TRIAL: NCT05813756
Title: Validation Study of the Coping, Motivation Ans Post-diagnosis Psychoeducation Program for Adults With Autism : a Randomized Controlled Trial
Brief Title: Validation Study of the Coping, Motivation and Post-diagnosis Psychoeducation Program for Adults With Autism
Acronym: CoMPPAA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Rouffach (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHR 10; 2022-A02489-34 (Other: COMITE DE PROTECTION DES PERSONNES SUD-EST VI)
Record Dates: First submitted 2023-03-20; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Psychoeducation; Autism; Self-determination; Adult
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental_Adults with Autism Spectrum Disorder (Experimental): post diagnostic psychoeducational intervention and filling of scale and questionnaire
  Interventions: Other: Post-diagnosctic psychoeducational intervention
- Adults with Autism Spectrum Disorder (No Intervention): Filling of scale and questionnaire.

INTERVENTIONS:
Other: Post-diagnosctic psychoeducational intervention — Participants are randomized to the intervention group. In this group, the participant receives 10 one-hour individual sessions of psychoeducational intervention, bi-monthly, with an evaluation at mid-term (T1:T0+~2.5 months), at the end of the intervention (T2 : T0+~5 months) and 3 months after the intervention (T3 : T0+~8 months). At the same time psychological questionnaires and scales will be completed
  Arms: Experimental_Adults with Autism Spectrum Disorder

SUMMARY:
The primary objective of the study is to evaluate the effectiveness of a post-diagnostic psychoeducational intervention in increasing the sense of self-efficacy of adults diagnosed with Autism Spectrum Disorder-Without associated Intellectual Disability

DETAILED DESCRIPTION:
Secondary objectives

The other objectives of this study are :

1. To evaluate the effectiveness of the intervention on self-esteem ;
2. To evaluate the effectiveness of the intervention on anxiety-depressive symptomatology ;
3. To evaluate the effectiveness of the intervention on the acceptance of the diagnosis ;
4. To evaluate the acceptance of the intervention.

Conduct of research The study will be offered to individuals diagnosed with autism spectrum disorder without associated intellectual developmental disabilities in adulthood.

After signing the consent form and verifying the eligibility criteria, participants will be randomized into the waiting list group or the intervention group.

In the intervention group : the participant will receive 10 one-hour individual sessions, bi-monthly, with an assessment at midterm (T1 : T0+~2.5 months), at the end of the intervention (T2 : T0 +~5 months) and 3 months after the intervention (T3 : T0 +~8 months).

In the waiting list group : the participant will receive the intervention at the exit of the research protocol (after T3).

At conclusion and at each visit, participants will complete questionnaires and scales defined in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged 18 years and older at the time of inclusion in the study
* Participant with a diagnosis of Autism Spectrum Disorder - Without associated Intellectual Disability (intelligence quotient > 80) made by a specialized 2nd (1) or 3rd (2) line team according to the recommendations of the Haute Autorité de la Santé (HAS)
* Diagnosis of Autism Spectrum Disorder - Without associated Intellectual Disability obtained in adulthood (≥ 18 years) within 15 months prior to inclusion
* Participant able to understand the objectives and risks of the research and having signed a consent to participate in the study
* Participant affiliated with a social security plan or beneficiary of such a plan

  1. Psychiatric teams (psychiatric services including medical-psychological centers), care networks specialized in the diagnosis and evaluation of autism or private practitioners coordinated by a physician.
  2. Professionals working in autism resource centers or hospitals for additional specialized medical advice, particularly in clinical genetics and medical imaging.

Exclusion Criteria:

* Participant not sufficiently available to participate in the intervention
* Participant in full hospitalization
* Participant co-morbid with schizophrenia or other psychotic disorder according to DSM-5 criteria
* Impossibility of giving the participant informed information (participant in an emergency or life-threatening situation, difficulties in understanding the participant, insufficient command of the French language)
* Participant under court protection or deprived of liberty by judicial or administrative decision
* Participant under guardianship or curatoship
* Diagnosed with Autism Spectrum Disorder - Without associated Intellectual Disability in childhood or adolescence or in a period of more than 15 months prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
General Self-Efficacy Scale | Change from inclusion result at 8 months
  It is a unidimensional scale that assesses beliefs in one's ability to achieve goals and to cope with and/or adapt to various situations that may arise in daily life. This measure consists of 10 items rated on a 4-point Likert scale (1= "not at all true" ; 4 = "completely true"). Overall scores range from 10 to 40, with higher scores indicating a greater sense of self-efficacy.

SECONDARY OUTCOMES:
Self-Esteem Scale | Through study completion , an average of 8 months
  This instrument, which assesses individuals' overall perception of their own worth, includes 10 items rated on a 4-point Likerts scale (1 = "strongly disagree", 4 = "strongly agree").
Depression Anxiety Stress Scale | Through study completion , an average of 8 months
  This instrument, which assesses psychological distress through indicators of stress and anxiety-depressive symptomatology (in the previous week), has been validated (in its English version) in an autistic population Without associated Intellectual Disability.
  This measure consists of 20 items rated on a 4-point Likert scale (1= "not at all" ; 4 = "all the time"). Overall scores range from 20 to 80, with higher scores indicating severe depression and anxiety
Acceptance and Action Questionnaire_Version 2 | Through study completion , an average of 8 months
  Questionnaire that specifically targets acceptance of Autism Spectrum Disorder diagnosis This measure consists of 7 items rated on a 7-point Likert scale (1= "never true" ; 7 = "always true"). Overall scores range from 7 to 49, with higher scores indicating a non-acceptance of the diagnosis
Social validity measures (in-house questionnaires) | Through study completion , an average of 8 months
  Acceptance of the intervention will be assessed by social validity measures that will take the form of a questionnaire developed in-house and including items on: expectations (visit 0) and satisfaction halfway through the intervention (visit 1) and (visit 2), use of strategies (visit 3) and knowledge about autism spectrum disorders.
  This measure consists of 10 items rated on a 4-point Likert scale (1= "completely disagree" ; 4 = "totally agree"). Overall scores range from 10 to 40, with higher scores indicating a high social validity.
qualitative data (semi-structured interviews) | Through study completion , an average of 8 months
  Acceptance of the intervention will be assessed by qualitative data collected through semi-structured interviews (visit 2 and visit 3: only for the "intervention" group with already defined themes).
  There is no score, then no minimum and maximum values (exchange in the form of organized notes).

CONTACTS AND LOCATIONS:
Overall Officials: ERIC BIZET, PhD, Principal Investigator — Autism Resource Center Colmar
Locations (1):
- Centre Hospitalier de Rouffach, Rouffach, France